CLINICAL TRIAL: NCT02162927
Title: The Effects of Six-day Dietary Nitrate Supplementation on Strength and Endurance Measurements in Male CrossFit Athletes
Brief Title: Dietary Nitrate Supplementation and Crossfit Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC2014
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Performance
Keywords: muscular strength; muscular endurance; muscular power; rowing; CrossFit; dietary nitrate
MeSH Terms: interventions — Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Potassium Nitrate (N) (Experimental): This involves 1 serving (2 pills) of potassium nitrate KNO3- (N) (8 mmols NO3-). The supplementation period is six days. This pill must be taken on an empty stomach (2-3 hours after eating) and must be taken about 2-3 hours before exercise.
  Interventions: Dietary Supplement: Dietary Nitrate
- Potassium Chloride (Placebo Comparator): This involves 1 serving (2 pills) of the nitrate-free placebo (PL) potassium chloride (8 mmol KCl) for a six-day supplementation period. This pill must be taken on an empty stomach (2-3 hours after eating) and must be taken about 2-3 hours before exercise.
  Interventions: Dietary Supplement: Potassium Chloride (placebo)

INTERVENTIONS:
Dietary Supplement: Dietary Nitrate — This pill must be taken on an empty stomach (2-3 hours after eating) and must be taken about 2-3 hours before exercise.
  Arms: Potassium Nitrate (N)
Dietary Supplement: Potassium Chloride (placebo) — This pill must be taken on an empty stomach (2-3 hours after eating) and must be taken about 2-3 hours before exercise.
  Arms: Potassium Chloride

SUMMARY:
In the past, dietary nitrate supplementation has been shown to have clinical benefits in the treatment of cardiovascular issues. More recently, however, the focus of nitrate supplementation has shifted to focus of human performance, and has shown to increase the time to exhaustion during maximal intensity exercise and lower the cost of oxygen consumption during submaximal intensity exercise. Acutely, nitrate supplementation in the form of beetroot juice has been shown to increase strength measurements, as well as increase the time to complete a 2000 meter rowing ergometer test. However, to the author's knowledge, there are no studies that link the relationship between multi-day nitrate supplementation and the rowing test or the nitrate's effect on strength when in the salt form. Additionally, to the author's knowledge, no evidence has been published which relates dietary nitrate supplementation and its effects on a CrossFit circuit workout.

Our central hypothesis is that six days of dietary nitrate supplementation will improve strength, endurance, a power more than a placebo in male CrossFit athletes.

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind, crossover study is to identify if dietary nitrate supplementation improves strength , endurance, and power measurements in male CrossFit athletes. Specifically, the strength measurements will be taken using isometric and isokinetic tests on the Biodex dynamometer. Endurance will be measured using time trials for a 2000 meter rowing test and the "Fran" CrossFit workout. Finally, power will be analyzed using the Wingate cycle test.

The treatment group will receive 1 serving of f potassium nitrate KNO3- (N) (8 mmols NO3-). The placebo group will receive 1 serving of the nitrate-free placebo (PL) potassium chloride (8 mmol KCl).

The participants will complete two three-day baseline testing, with a six-day supplementation period following each round of baseline testing. Following the first six-day supplementation period, there will be a 10 day washout period before the second baseline testing begins.

ELIGIBILITY:
Inclusion Criteria:

* College-aged male CrossFit between the ages of 20 and 35 years (yr), a peak maximum oxygen uptake (VO2peak) of at least 50 ml/kg/min will be recruited to participate in this study.

Exclusion Criteria:

* Having any thyroid and/or kidney diseases that could affect NO synthesis and/or metabolism, any illness, smoking, taking other medications, injured, not well-trained (as noted by the VO2peak), consuming any other supplements at the time of the study except protein or multivitamin, allergic to any component of the supplement, including tree nuts, in case of potential packaging mixing and contamination. Women and children as well are excluded.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Muscular Strength | During 1 month of study
  Muscular Strength will be tested using the isometric and isokinetic strength tests.
Muscular Endurance | 1 month
  Endurance will be tested using the 2000 meter rowing ergometer test and CrossFit circuit known as "Fran".
Muscular Power | 1 month
  Power will be measured using the Wingate cycle test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ormsbee, PhD, Principal Investigator — Florida State University; Samuel J Kramer, BS, Study Director — Florida State University
Locations (2):
- United States (2):
  - CrossFit Blackbox, Tallahassee, Florida
  - Florida State University, Tallahassee, Florida